CLINICAL TRIAL: NCT01681732
Title: A Pilot Study of Personalized Medicine for Pediatric Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 38403
Record Dates: First submitted 2012-09-05; First posted 2012-09-10 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Asthma
Keywords: Asthma; child; pediatric
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Personalized Care Plan (Experimental): A personalized plan based on baseline clinic visit data
  Interventions: Other: Personalized Care Plan
- Control (Active Comparator): This arm will be standard care
  Interventions: Other: Control Standard Care

INTERVENTIONS:
Other: Personalized Care Plan — We will develop a personalized plan based on info collected in the primary visit
  Arms: Personalized Care Plan
Other: Control Standard Care — This is the standard care arm
  Arms: Control

SUMMARY:
A pilot study to test the feasibility of a personalized asthma care intervention.

DETAILED DESCRIPTION:
There are two arms in this study. The control arm of the trial will involve the current standard primary care asthma management, and the intervention arm will involve personalized asthma management.

Inclusion criteria include: 1) child age 6-17 years, 2) doctor diagnosed asthma, 3) at least one asthma exacerbation in the previous year. Children with other coexistent pulmonary diseases such as chronic lung disease and cystic fibrosis will be excluded.

The period of participation will be three months for each participant. After screening, each participant will have an initial clinic visit. During this baseline visit, the investigators will collect DNA by taking a saliva sample, the investigators will conduct spirometry, and the investigators will survey the families regarding household level environmental exposures, demographics, and other key variables. The participant will be randomly assigned to a study arm at the end of the baseline visit. The data gathered at the baseline visit will be used to develop a management plan. The investigators will mail a plan to the participant and the primary care provider within a couple weeks of the baseline visit. The investigators will then discuss the plan with the participant via phone. Both groups will receive a plan which MAY be used to guide asthma care. Sample letters follow the protocol. The intervention group will receive basic information on the skin testing, genetic testing, and spirometry. The control group will not receive the genetic information. The control arm will receive the genetic information at the end of the study follow up.

After the baseline visit, the participants will receive a monthly phone call for two months to conduct a survey to assess our study outcomes and covariates. At the 3rd month participants will return to the GCRC for a final clinic visit. During the final visit the investigators will conduct our survey and spirometry and request permission for medical record release.

ELIGIBILITY:
Inclusion Criteria:

* age 6-17 years
* doctor diagnosed asthma -at least one asthma exacerbation in the previous year. -

Exclusion Criteria:

-Children with other coexistent pulmonary diseases such as chronic lung disease and cystic fibrosis will be excluded.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2012-09; Primary Completion 2014-08-29 (Actual); Study Completion 2014-08-29 (Actual)

PRIMARY OUTCOMES:
number of symptom free days over the course of the study | 3 months
  measured as the number of days during the 2 weeks before the follow-up interview with no asthma symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Adam Spanier, MD, PhD, MPH, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Children's Hospital, Hersey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No